CLINICAL TRIAL: NCT06293326
Title: An Open Label, Single Center, Randomized, Two-way Crossover Parallel Group, Trial to Assess the Mechanism of Action of a Bi-layer Swallowable Tablet (Immediate Release and Sustained Release) Containing Calcium Carbonate Antacid in an Overnight and Day Application as Compared With a Standard, Non-layered (Immediate Release) Calcium Carbonate Swallow Tablet in Fed Healthy Male Participants.
Brief Title: A First-in-Human Study to Learn How Well a Bi-Layer Calcium Carbonate Antacid Tablet Works Compared to a Standard, Non-Layered Calcium Carbonate Tablet in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22553
Record Dates: First submitted 2024-02-16; First posted 2024-03-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Heartburn; Indigestion; Stomach Acid Related Symptoms; Nocturnal Stomach Acid Related Symptoms; Healthy Volunteers
MeSH Terms: conditions — Heartburn; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night-time sequence (Experimental): The night-time treatment sequence consists of two Treatment periods (Period 1 and Period 2) with each period consisting of a single dose of Investigational Medicinal Product (IMP). The two Treatment periods are separated by a least 6-8-day wash-out phase between IMP administration in Period 1 and 2.
  Interventions: Drug: bi-layer calcium carbonate tablet (BAY1180654); Drug: Immediate release calcium carbonate tablet (BAY1180654)
- Day-time sequence (Experimental): The day-time treatment sequence consists of two Treatment periods (Period 1 and Period 2) with each period consisting of a single dose of IMP. The two Treatment periods are separated by a least 6-8-day wash-out phase between IMP administration in Period 1 and 2.
  Interventions: Drug: bi-layer calcium carbonate tablet (BAY1180654); Drug: Immediate release calcium carbonate tablet (BAY1180654)

INTERVENTIONS:
Drug: bi-layer calcium carbonate tablet (BAY1180654) — Singal dose; two tablets; administered 1-2 hours post standardized meal depending on day or night dosing.
Drug: Immediate release calcium carbonate tablet (BAY1180654) — Singal dose; two tablets; administered 1-2 hours post standardized meal depending on day or night dosing.

SUMMARY:
Researchers are looking for a better way to treat people who have heartburn, indigestion, and problems due to excessive stomach acid. These are common problems which can affect daily life and disturb sleep during the night-time. Heartburn is the burning sensation or pain in the chest which occurs when stomach acid rises up in the food pipe (esophagus).

Calcium carbonate tablets are used to treat heartburn, indigestion, and related digestive problems. Calcium carbonate works by neutralizing the excess acid in the stomach. The study treatment is a new bi-layer calcium carbonate tablet that has two layers. One layer quickly releases calcium carbonate aimed to provide quick relief (called immediate release) while the other layer releases calcium carbonate slowly to make the relief last longer (called sustained release).

In this study, bi-layer calcium carbonate tablets will be given to healthy men for the first time. This study will provide information on how the new bi-layer tablet works inside the body.

The main purpose of this study is to learn about how the new bi-layer calcium carbonate tablet changes the average acidity levels (measured using pH) compared to the standard calcium carbonate tablet during the night-time.

For this, researchers will measure the acidity levels in the upper part of the stomach at regular intervals during the night-time.

The participants will be randomly (by chance) assigned to one of two treatment groups:

Participants in the first group will take the treatments at night.

Participants in the second group will take the treatments during the day.

All participants in both groups will take 2 bi-layer tablets and 2 standard tablets after a meal with a gap of 6 to 8 days between treatments. However, in each group, half the participants will receive the bi-layer tablets first while the other half will receive the standard tablets first.

Each participant will be in the study for around 52 days with up to 4 visits to the study site. This includes:

1. visit about 28 days before the treatment starts during which the doctors will confirm that the participant can take part in the study
2. visits for treatment with a gap of 6-8 days between each treatment, and

1 visit 7 to 14 days after the treatment ends during which the doctors will monitor the participants' health.

During the study, the doctors and their study team will:

check participants' overall health by performing tests such as blood and urine tests, and check heart health using an electrocardiogram (ECG)

take images of the stomach at different times after taking the treatment

measure acidity level (pH) using a device called pH probe that is inserted into the upper part of the stomach

ask the participants questions about how easy it is to take the study treatment

ask the participants what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think it is related to the study treatment, or not.

As this study is conducted in healthy men who will not gain any benefit from this treatment, access to the study treatment after the study is not planned.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Participant must be 18 to ≤65 years of age inclusive, at the time of signing the informed consent.
* Participants must have a verified diagnosis of "healthy": the results of the standard clinical, laboratory, and instrumental examinations are within the normal range (limits of reference range). The Investigator can interpret individual findings based on the participant's age, physical state and level of fitness. Participants with readings marginally outside the normal range may be included in the study if, in the Investigator's opinion, these are not clinically significant (NCS); this decision will be documented in the Case Report Form (CRF).
* Results of safety laboratory tests are within normal range (limits of reference range).
* Non-smokers or passive smokers exposed to smoke in an enclosed room for less than 4 h per week.
* Body mass index (BMI) within the range 18.5 to ≤30 kg/m2 (inclusive).
* Unless participant has had bilateral orchidectomy or a vasectomy (with confirmed sterility), must be abstinent from penile-vaginal intercourse for the duration of the study and agree to remain abstinent for 90 days after the last dose of IMP, OR agree to use a condom during each episode of penile-vaginal intercourse, in addition to their partner (if a person who could become pregnant) using a highly effective form of contraception as described in protocol.
* Participant has given written informed consent to participate in the trial prior to admission to the trial as described in the protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Be willing and able to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the protocol.

Exclusion Criteria:

* A history of physical or psychiatric diseases (e.g., diabetes, hypothyroidism and other metabolic diseases, renal disease).
* Recent unexplained significant weight loss (6-7 kg) in the last 6 months.
* A history or current symptoms of Zollinger-Ellison syndrome, gastric carcinoma, peptic ulcer disease, pernicious anaemia, Barrett's oesophagus or systemic sclerosis.
* Meal-induced heartburn of severe severity, historically and -
* Use of any H2-receptor antagonist and/or PPI within one week prior to Screening.
* History and currently prescribed medication for treatment of heartburn associated with increased acidity, reflux esophagitis, and peptic ulcers.
* Current or history of drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Gastric pH levels as measured and recorded with tip of pH probe in gastric fundus. | During night-time on Day 1

SECONDARY OUTCOMES:
Gastric pH levels as measured and recorded with tip of pH probe in gastric fundus. | During daytime on Day 1
Percentage of total time gastric pH is above pH 3.5 from time of dosing until 8h post-dose during night-time comparing the bi-layer tablet and standard comparator | Up to 8 hours post-dose during night-time
Percentage of total time gastric pH is above pH 3.5 from time of dosing until 6h post-dose during daytime comparing the bi-layer tablet and standard comparator. | Up to 6 hours post-dose during daytime
Change in mean gastric pH | During night-time and daytime on Day 1
Gastrointestinal tract location using scintigraphic images. | During night-time and daytime on Day 1
Initial radiolabel release time, using scintigraphic images | During night-time and daytime on Day 1
Disintegration rate (t50%) of each formulation will be determined quantitatively via analysis of scintigraphic images. | During night-time and daytime on Day 1
Complete radiolabel release time, using scintigraphic images | During night-time and daytime on Day 1
Gastric emptying kinetics of the dispersed radiolabeled material (t50% and t90%) of each formulation will be determined quantitatively via analysis of the scintigraphic images. | During night-time and daytime on Day 1
Participant questionnaire | On Day 1
  The following questions will be asked:
  PERCEPTIONS Focusing on the sensory experience you have had from the tablet; please indicate how much you agree/disagree with each of the following statements?
  * This tablet feels like is easy to swallow
  * This tablet is pleasant to use

CONTACTS AND LOCATIONS:
Locations (1):
- BDD Pharma Bio-imaging Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22553